CLINICAL TRIAL: NCT05619055
Title: The Role and Mechanism of Intestinal Dysbacteriosis Impairing the Intestinal Mucosal Barrier in the Pathogenesis of Necrotizing Enterocolitis in Premature Infants
Brief Title: The Intestinal Dysbacteriosis in the Pathogenesis of Necrotizing Enterocolitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zuohui Zhao (Other)
Responsible Party: Sponsor-Investigator, Zuohui Zhao, Associate professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2022(018)
Record Dates: First submitted 2022-11-02; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Necrotizing Enterocolitis of Newborn
Keywords: Necrotizing Enterocolitis; intestinal flora
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neonate with necrotizing enterocolitis: premature infants diagnosed as necrotizing enterocolitis
  Interventions: Other: Routine treatment
- neonate without necrotizing enterocolitis: premature infants without necrotizing enterocolitis
  Interventions: Other: Routine treatment

INTERVENTIONS:
Other: Routine treatment — Antibiotics, intravenous fluids and symptomatic supportive treatment.

SUMMARY:
Study Description

The goal of this observational study is to detect intestinal flora and the metabolic products in premature infants diagnosed as necrotizing enterocolitis. The main questions it aims to answer are:

* 1. Whether there is intestinal flora in the stool of premature infants.
* 2. Are there dysregulated intestinal flora and their metabolic products in premature infants diagnosed as necrotizing enterocolitis.
* 3. The detailed role and underlying mechanism of the intestinal dysbacteriosis and the metabolic products in premature infants diagnosed as necrotizing enterocolitis.

Participants, premature infants diagnosed as necrotizing enterocolitis (NEC group), will be asked to collect stool (usually 2 times) for intestinal flora analysis.

If there is a comparison group: Researchers will compare premature infants without necrotizing enterocolitis (control group) to see if their intestinal flora and the metabolic products also changed as their NEC counterparts.

DETAILED DESCRIPTION:
When the patients is hospitalized in neonatology, we screen the premature infants according to the selection criteria and exclusion criteria. After sighed the informed consent, they are classified into two groups: premature infants diagnosed as necrotizing enterocolitis (NEC group) and premature infants without necrotizing enterocolitis (control group). Their stool and blood (usually 2 times ) are collected for intestinal flora and FABP (including L-FABP and I-FABP) analysis, respectively.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Necrotizing Enterocolitis,
* gestational age <37 weeks,
* body weight 1,000-2,500 g,
* postnatal Apgar score ≥7,
* initial oral feeding tolerance.

Exclusion Criteria:

* serious hereditary or other serious diseases, such as heart, lung and abdominal malformations ,
* early or late onset septicemia,
* early use of antibiotics in the newborn,
* serious adverse reactions caused by probiotics.

Ages: 5 Days to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Hospitalized children in Neonatology
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-11-05 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
intestinal flora | up to 4 weeks
  the intestinal flora in the stool using 16S ribosomal RNA(rRNA) gene sequencing
short-chain fatty acids | up to 4 weeks
  short-chain fatty acids, the metabolic products of intestinal flora, in the stool using 16S rRNA gene sequencing
neurotransmitters | up to 4 weeks
  neurotransmitters, the metabolic products of intestinal flora, in the stool using 16S rRNA gene sequencing
lipopolysaccharide | up to 4 weeks
  lipopolysaccharide, a metabolic product of intestinal flora, in the stool using 16S rRNA gene sequencing
L-FABP | up to 4 weeks
  L-FABP, the injury marker of intestinal mucosa, in the blood
I-FABP | up to 4 weeks
  I-FABP, the injury marker of intestinal mucosa, in the blood
hospital stay | up to 4 weeks
  one vital clinical outcome of the premature infants

SECONDARY OUTCOMES:
X-ray | up to 4 weeks
  one important clinical imaging data of the premature infants
complete blood count | up to 4 weeks
  complete blood count, one vital laboratory test of the premature infants
c-reactive protein | up to 4 weeks
  c-reactive protein, one vital laboratory test of the premature infants
procalcitonin | up to 4 weeks
  procalcitonin, one vital laboratory test of the premature infants

CONTACTS AND LOCATIONS:
Overall Officials: Zuohui Zhao, Dr, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided
The clinical data to collect for individual participant is not public for the time being.